CLINICAL TRIAL: NCT01254643
Title: A Phase III Open-label, Safety, Tolerability and Immunogenicity Study of a 9-Valent Human Papillomavirus (HPV) L1 Virus-Like Particle (VLP) Vaccine Administered to 9- to 15-Year-Old Japanese Preadolescent and Adolescent Girls
Brief Title: A Study of the Safety, Tolerability, and Immunogenicity of a 9-valent Human Papillomavirus Vaccine ([9vHPV]; V503) Administered to 9- to 15-Year-Old Japanese Girls (V503-008).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V503-008
Record Dates: First submitted 2010-12-03; First posted 2010-12-06 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2018-11-28 (Actual); Status verified 2018-10

CONDITIONS: Papillomavirus Infections
Keywords: Papillomavirus vaccines; Uterine cervical cancer; Human Papilloma Virus infections
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Enrolled (Experimental): 9-valent human papillomavirus (9vHPV) L1 VLP vaccine (V503), 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6.
  Interventions: Biological: V503

INTERVENTIONS:
Biological: V503 — V503 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6

SUMMARY:
This study will evaluate the safety, tolerability, and immunogenicity of V503 in Japanese girls between the ages of 9 and 15 and will determine whether V503 induces an acceptable immune response to all human papillomavirus (HPV) strains contained in the vaccine. The success criterion for the primary analysis requires that point estimates for seroconversion rate be greater than 90% for all 9 HPV types.

ELIGIBILITY:
Inclusion Criteria:

* Participant is in good physical health-
* Participant's parent/legal guardian is able to read, understand, and complete the vaccine report card
* Participant's parent/legal guardian agrees to provide a phone number for follow-up purposes
* Participant is not sexually active and does not plan to become sexually active during the time from Day 1 to Month 7 of the study

Exclusion Criteria:

* Participant has a history of severe allergic reaction that required medical intervention
* Participant has thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injection
* Participant is pregnant
* Participant intends to donate blood during the time from Day 1 to Month 7 of the study
* Participant is immunocompromised or has been diagnosed as having a congenital or acquired immunodeficiency, human immunodeficiency virus (HIV) infection, lymphoma, leukemia, systemic lupus erythematosus, rheumatoid arthritis, juvenile rheumatoid arthritis, inflammatory bowel disease, or other autoimmune condition.
* Participant has had a splenectomy
* Participant has received any of the following immunosuppressive therapies in the year prior to enrollment: radiation therapy, cyclophosphamide, azathioprine, methotrexate, any chemotherapy, cyclosporin, leflunomide (Arava), tumor necrosis factor alpha (TNF-α) antagonists, monoclonal antibody therapies, antilymphocyte sera, or other therapy known to interfere with the immune response.
* Participant has received any immune globulin product or blood-derived product in the three months prior to the Day 1 vaccination, or plans to receive any such product through Month 7 of the study
* Participant has received any inactivated vaccines within 14 days of the Day 1 vaccination or any live vaccines within 28 days of the Day 1 vaccination
* Participant has received a marketed HPV vaccine or has participated in an HPV vaccine clinical trial
* Participant has had a fever (oral temperature ≥37.8°C) within 24 hours of the Day 1 vaccination
* Participant has a history of a positive test for HPV or history of genital warts

Ages: 9 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2011-01-12 (Actual); Primary Completion 2013-08-10 (Actual); Study Completion 2013-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Iwata S, Murata S, Rong Han S, Wakana A, Sawata M, Tanaka Y. Safety and Immunogenicity of a 9-Valent Human Papillomavirus Vaccine Administered to 9- to 15-Year-Old Japanese Girls. Jpn J Infect Dis. 2017 Jul 24;70(4):368-373. doi: 10.7883/yoken.JJID.2016.299. Epub 2016 Dec 22. PMID 28003597
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=V503-008&kw=V503-008&tab=access

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Enrolled
Started | 100
Vaccination 1 | 100
Vaccination 2 | 99
Vaccination 3 | 99
Completed | 99
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled: 9-valent human papillomavirus (9vHPV) L1 VLP vaccine, 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6.
Arm/Group | All Enrolled
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.7 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Seroconvert to Each of the HPV Types Contained in the Vaccine
Description: Serum antibody titers for HPV virus-like particles (VLPs), Types 6, 11, 16, 18, 31, 33, 45, 52 and 58 were determined 4 weeks post-vaccination 3 using competitive luminex immunoassay (cLIA). The serostatus cutoffs (milli Merck U/mL) for HPV types were as follows: HPV Type 6: ≥30, HPV Type 11: ≥16; HPV Type 16: ≥20, HPV Type 18: ≥24, HPV Type 31: ≥10, HPV Type 33: ≥8, HPV Type 45: ≥8, HPV Type 52: ≥8, and HPV Type 58: ≥8.
Time Frame: 4 weeks post-vaccination 3 (Month 7)
Population: Participants who received all 3 vaccinations and met criteria for Per Protocol Immunogenicity (PPI) Population (not a general protocol violator, received all vaccinations within acceptable day ranges, seronegative at Day 1 for HPV type(s), and had a Month 7 serum sample collected within an acceptable day range) for at least 1 of the 9 HPV types.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 99
Percentage of Participants
  Anti-HPV 6 (n=97) | 100 [96.3 to 100]
  Anti-HPV 11 (n=97) | 100 [96.3 to 100]
  Anti-HPV 16 (n=99) | 100 [96.3 to 100]
  Anti-HPV 18 (n=98) | 100 [96.3 to 100]
  Anti-HPV 31 (n=97) | 100 [96.3 to 100]
  Anti-HPV 33 (n=98) | 100 [96.3 to 100]
  Anti-HPV 45 (n=99) | 100 [96.3 to 100]
  Anti-HPV 52 (n=99) | 100 [96.3 to 100]
  Anti-HPV 58 (n=95) | 100 [96.2 to 100]

2. Primary Outcome: Percentage of Participants With an Injection-site Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the vaccine. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an AE. AEs such as redness, swelling, and pain/tenderness/soreness at the injection site were recorded.
Time Frame: up to 5 days after any vaccination
Population: Safety Population, which consisted of all participants who received at least one vaccination and had available follow-up data.
Measure: Number; unit: Percentage of Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 100
Percentage of Participants | 95.0

3. Primary Outcome: Percentage of Participants With a Non-Injection Site (Systemic) AE
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the vaccine. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an AE. Systemic AEs were those not categorized as injection-site AEs.
Time Frame: up to 15 days after any vaccination
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 100
Percentage of Participants | 35.0

4. Primary Outcome: Percentage of Participants With a Vaccine-related AE
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the vaccine. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an AE. Adverse experience that is judged by the Investigator to be "definitely related," "probably related," or "possibly related" to the study drug is defined as a vaccine-related AE.
Time Frame: up to 15 days after any vaccination
Population: Safety Population, which consists of all participants who received at least one vaccination and had available follow-up data.
Measure: Number; unit: Percentage of Participants
Arm/Group | All Enrolled
Number analyzed (Participants) | 100
Percentage of Participants | 96.0

5. Secondary Outcome: Geometric Mean Titers (GMTs) for Each of the HPV Types Contained in the Vaccine
Description: Serum antibody titers for HPV virus-like particles (VLPs), Types 6, 11, 16, 18, 31, 33, 45, 52 and 58 were determined 4 weeks post-vaccination 3 using cLIA. Titers are reported in milli Merck Units/mL.
Time Frame: 4 weeks post-vaccination 3 (Month 7)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: milli Merck units/mL
Arm/Group | All Enrolled
Number analyzed (Participants) | 99
milli Merck units/mL
  Anti-HPV 6 (n=97) | 1836.5 [1597.7 to 2111.0]
  Anti-HPV 11 (n=97) | 1331.3 [1135.0 to 1561.4]
  Anti-HPV 16 (n=99) | 6823.6 [5907.9 to 7881.2]
  Anti-HPV 18 (n=98) | 2159.9 [1803.8 to 2586.3]
  Anti-HPV 31 (n=97) | 2052.5 [1735.9 to 2426.8]
  Anti-HPV 33 (n=98) | 994.8 [857.2 to 1154.4]
  Anti-HPV 45 (n=99) | 811.0 [679.7 to 967.6]
  Anti-HPV 52 (n=99) | 1069.1 [908.4 to 1258.4]
  Anti-HPV 58 (n=95) | 1488.2 [1285.0 to 1723.4]

ADVERSE EVENTS:
Time Frame: Up to 5 days after any vaccination (Non-serious injection site AEs); up to 15 days after any vaccination (Serious AEs and Non-serious non-injection site AEs) and up to 30 months (Any death and serious drug-related AEs)
Description: Safety Population, which consisted of all participants who received at least one vaccination and had available follow-up data.
Arm/Group | All Enrolled
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 96/100
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled (N=100)
Injection site erythema (General disorders) | 33 (57)
Injection site pain (General disorders) | 93 (241)
Injection site swelling (General disorders) | 42 (67)
Pyrexia (General disorders) | 6 (6)
Nasopharyngitis (Infections and infestations) | 9 (9)
Headache (Nervous system disorders) | 8 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines